CLINICAL TRIAL: NCT00631397
Title: A Preliminary Study of Bone Density Measurements in Neonates Using the Sunlight Omnisense 7000P Ultrasound Bone Sonometer
Brief Title: A Preliminary Study of Bone Density in Neonates
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 5974; University of South Florida; Grant
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2007-03

CONDITIONS: Osteopenia Of Prematurity
Keywords: weakening of the bones
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Measuring proteins in the blood plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Premature Infants: Premature Infants weighing less than 1500 gms
  Interventions: Device: Ultrasound machine

INTERVENTIONS:
Device: Ultrasound machine — Weekly Bone Density measurements using the Sonometer
  Other Names: Omnisense 7000P Ultrasound Bone Sonometer

SUMMARY:
The study is to measure how dense or solid the infant's bones are using a new ultrasound machine and how that density changes over time.

DETAILED DESCRIPTION:
premature infants weighing less than 1500 gms and less than 33 weeks gestation are eligible for the study

ELIGIBILITY:
Inclusion Criteria:

* premature infants born less than 33 weeks, weighing less than 1500 gms

Exclusion Criteria:

* congenital anomalies weight greater than 1500 gms

Ages: 24 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature Infants In the Neonatal Intensive Care Unit
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Develop ways to prevent and treat Osteopenia of Prematurity | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Terri L Ashmeade, M.D., Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital/University of South Florida, Tampa, Florida, United States